CLINICAL TRIAL: NCT04060693
Title: Device Accuracy of Non-invasive Glucose Measurements in Ethnic Skin
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Miscommunication with the CRO that was hired to help with the regulatory submission process
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RSP 18
Record Dates: First submitted 2018-10-12; First posted 2019-08-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus
Keywords: Non-invasive glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Open, non-randomized comparison study between device and blood references with diabetic patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protocol 1 (Experimental): The subjects enrolled in this protocol will dedicate 30 days of home-based measurement, scheduled within a 40 days' time frame. For reference measurements, subjects will be equipped with a BG-meter (Contour Next One, Ascenia). Optical measurements are collected with the IMD. Each day of measurements consists of four sessions each comprising two capillary blood glucose measurement with a BG-meter and two IMD measurements. IMD measurements will be performed within 3 minutes after the BG measurement using the thenar of the right hand of the subject.
  Interventions: Device: P0.5

INTERVENTIONS:
Device: P0.5 — Investigational Medical Device collecting spectral raman data from tissue.

SUMMARY:
This clinical study has been launched to collect spectral raman data paired with validated glucose reference values in private homes of subjects.

DETAILED DESCRIPTION:
The subjects enrolled in this protocol will dedicate 30 days of home-based measurement, scheduled within a 40 days' time frame. For reference measurements, subjects will be equipped with a blood glucose meter (Contour Next One, Ascenia). Optical measurements are collected with the investigational medical device. Each day of measurements consists of four sessions each comprising two capillary blood glucose measurement with a blood glucose meter and two investigational medical device measurements.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years of age.
* Have a diagnosis of diabetes mellitus.
* Distribution of skin phototype: 50-70 % of enrolled subjects phototype IV, 20-40 % of enrolled subjects phototype III, 5-15 % of enrolled subjects phototype II, 5-15 % of enrolled subjects phototype I.
* Be willing to perform a minimum of 8 finger sticks per day during the study.
* Be willing to perform a minimum of 8 optical measurements per day during the study.
* Be willing to provide written signed and dated informed consent.

Exclusion Criteria:

* Breastfeeding, pregnant, attempting to conceive or not willing and able to practice birth control during the study execution (applicable to female subjects only).
* Subjects not able to understand and read English.
* Inability to comply with the study procedures as described by the study protocol, according to the opinion of the investigator.
* Subject is not able to hold hand/arm steadily (including tremors and Parkinson's Disease).
* Diagnosed with cardiovascular diseases.
* Reduced circulation in right hand evaluated by Allen's test.
* Subjects receiving anticoagulants, active cancer treatment, tetracyclines and other medication/topical agents increasing photosensitivity.
* Radiotherapy for the past six months.
* Extensive skin changes, tattoos or diseases on probe application site (thenar) that could interfere with the accuracy of the interstitial glucose measurements.
* Known allergy to medical grade alcohol used to clean the skin.
* Systemic or topical administration of glucocorticoids for the past 7 days and under investigation.
* Subjects undergoing dialysis treatment.
* Concomitant medical condition which could present a risk to the safety or welfare of the subject or study staff.
* Medical history or any condition that may, in the opinion of the investigator, compromise subject's ability to participate.
* Subjects currently enrolled in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Measurement accuracy of IMD | 8 months
  Accuracy of measurements performed on the IMD will be evaluated by data from subjects. Data will be analyzed by Mean Absolute Relative Difference (MARD).

SECONDARY OUTCOMES:
Safety evaluation: paucity of adverse events | 8 months
  Safety of the IMD will be evaluated in a descriptive manner by the paucity of adverse events reported during the clinical study.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Rare Disease ITM, Heritage Building (Queen Elizabeth Hospital Birmingham), Birmingham, Edgbaston, United Kingdom

IPD SHARING:
Plan to Share IPD: No